CLINICAL TRIAL: NCT01526707
Title: The Use of FKBP51 in the Identification of Non-adherence to Inhaled Corticosteroids in Difficult Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liam Heaney (Other)
Collaborators: Northern Ireland Chest Heart and Stroke (Other)
Responsible Party: Sponsor-Investigator, Liam Heaney, Consultant Physician, Belfast Health and Social Care Trust
Organization: Belfast Health and Social Care Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 10174LH-AS; 10174LH-AS (Other: Belfast Health & Social Care Trust); 11/NI/0015 (Other: Regional Ethics Committee Northern Ireland)
Record Dates: First submitted 2012-02-01; First posted 2012-02-06 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Asthma
Keywords: To identify changes in FKBP51 expression with inhaled steroid treatment in asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- inhaled steroid (Experimental): inhaled steroid treatment for 7 days
  Interventions: Drug: inhaled steroid

INTERVENTIONS:
Drug: inhaled steroid — inhaled budesonide for 7 days

SUMMARY:
Approximately 5-10% of people with asthma do not respond to to standard therapy and are referred to as having difficult asthma. Evidence shows that this poor response is not always related to asthma severity and non-adherence to treatment is recognized as a common underlying problem, in 35% of these patients. Recognising non-adherence in the clinic is problematic as there is no straightforward objective test to identify it.

Previous studies have demonstrated up-regulation of FKBP51 gene expression following treatment with steroids, making it a potential biomarker of steroid exposure. It is therefore also a potential biomarker of non-adherence to inhaled corticosteroid therapy. The investigators plan to assess the feasibility of distinguishing non-adherent subjects who are by omission steroid naïve from adherent subjects, steroid exposed subjects using FKBP51 gene expression in sputum and throat swabs.

To do this the investigators will obtain throat swab and sputum samples from healthy volunteers, steroid naïve asthmatics and adherent asthmatics on high dose ICS to assess if FKBP51 gene expression is comparable in each group.

The investigators will then compare the FKBP51 gene expression response to directly observed inhaled steroid therapy in steroid naïve, non-adherent and adherent asthmatics. This will identify if the response in gene expression distinguishes steroid exposed (adherent) from steroid naïve (non-adherent) patients.

Identifying non-adherence will benefit patients by enabling appropriate tailored management for non-adherence to enhance treatment effectiveness. It will also identify patients with therapy resistant asthma who have an unmet need and may benefit from expensive novel therapies such as Omalizumab.

ELIGIBILITY:
Inclusion Criteria:

This pilot study will investigate the following groups (n=10 per group):

1. Healthy volunteers.
2. Steroid naïve asthmatics.
3. Refractory asthmatics adherent to high dose inhaled steroids.
4. Non-adherent asthmatics.

Inclusion Criteria

For inclusion into this study all participants must:

* be 16 years old or older
* give written informed consent

Healthy volunteers must:

* be in good general health as determined by past medical history and physical.
* have no other significant medical history and specifically no prior history of asthma or persistent respiratory symptoms.
* normal spirometry.

Steroid naïve subjects

* have a diagnosis of asthma
* receiving treatment at Step 1 BTS/SIGN Guidelines i.e. no inhaled steroid

Non-adherent subjects must

* have a diagnosis of asthma
* be non-adherent to ICS as determined by ICS prescription filling of </=50% in the previous 6 months

Refractory asthmatic adherent subjects must:

* have a diagnosis of asthma receiving high dose ICS treatment (beclomethasone equivalent dose > 1000 µg per day)
* be adherent to ICS as determined by ICS prescription filling >75% in the previous 6 months

Exclusion Criteria:

Participants who fulfill the following criteria will be excluded from study entry:

* Current smoker,
* Pregnant or lactating,
* Other significant respiratory disease
* Previous allergic reaction or known hypersensitivity to budesonide or any corticosteroid

Healthy volunteers will be excluded if they have / are :

* any significant medical history which the principal investigator (PI) deems appropriate to be excluded from the healthy control group
* obstructive lung function
* taking any medication
* a current or history of drug or alcohol abuse
* any significant illness during the screening period preceding entry into the study

Steroid naïve / Non-adherent asthmatics will be excluded if they have:

* commenced or increase of oral corticosteroids in the previous 28 days
* a concurrent asthma exacerbation

Refractory / Adherent asthmatics will be excluded if they have:

* commenced or increased of oral corticosteroids in the previous 28 days
* a concurrent asthma exacerbation

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in FKBP51 gene expression | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Belfast City Hospital, Belfast, United Kingdom